CLINICAL TRIAL: NCT05943288
Title: Safety and Efficacy of the Olympus Endoscopy Computer-Aided Detection (CADe) System in Detection of Colorectal Neoplasia's During Real-time Colonoscopy: A European Prospective, Multicenter, Randomized Controlled Trial (EuroCADe)
Brief Title: Safety and Efficacy of the Olympus CADe System in Real-time Colonoscopy
Acronym: EuroCADe
Status: Completed | Type: Observational
Sponsor: Olympus Europe SE & Co. KG (Industry)
Collaborators: Cromsource (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP2021-AI (OEKG)-01
Record Dates: First submitted 2023-06-07; First posted 2023-07-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer
Keywords: AI (Artificial Intelligence); CADe (Endoscopy Computer Aided Detection)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CADe +: Olympus Endoscopy Computer-Aided Detection (CADe) system
  Interventions: Device: OIP-1
- CADe -: Standard of Care Endoscopy (HD Whitelight)

INTERVENTIONS:
Device: OIP-1 — Olympus Endoscopy Computer-Aided Detection (CADe) system
  Groups: CADe +

SUMMARY:
This is a prospective, multicenter, randomized Trial to assess the safety and efficacy of the Olympus Endoscopy Computer-Aided Detection (CADe) system, OIP-1, in the detection of colorectal neoplasia's during real-time colonoscopy. The aim of this system is to improve physician performance in the detection of potential mucosal abnormalities during colonoscopy performed for primary Colorectal Cancer screening or postpolypectomy surveillance.

DETAILED DESCRIPTION:
This Study aims to provide insight into whether the application of Artificial Intelligence (Olympus Endoscopy Computer-Aided Detection (CADe) system) increases the detection rate of adenomatous polyps in screening and / or surveillance colonoscopy procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. 45-80 years
3. Undergoing colonoscopy for primary CRC screening or postpolypectomy surveillance

Exclusion Criteria:

1. Lack of informed written consent
2. History of CRC or inflammatory bowel disease or polyposis syndrome / familial adenomatous polyposis coli (FAP)
3. Prior failed colonoscopy

   * multiple historic prior failed colonoscopy due to poor bowel preparation OR
   * a single prior failed colonoscopy due to reasons other than poor bowel preparation
4. Biopsy/anesthesia/sedation contraindications
5. History of radio- and/or chemotherapy
6. Concurrent participation in another competing clinical study

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing a colonoscopy
Sampling Method: Probability Sample
Enrollment: 850 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Adenoma Detection Rate (ADR) | During procedure
  Proportion of patients with at least one histologically confirmed adenoma (including advanced adenomas) or carcinoma in the CADe assisted colonoscopy (CADe+ arm) versus conventional colonoscopy without CAD (CADe- arm).
Positive Predictive Value (PPV) | During procedure
  Number of histologically confirmed polyps (i.e. adenomas, SSLs, or large (>10mm) hyperplastic polyps divided by the total number of resections.

SECONDARY OUTCOMES:
Adenoma Per Colonoscopy (APC) | During procedure
  Number of histologically proven adenomas (including advanced adenomas) or carcinomas divided by the total number of colonoscopies
Total Procedure Time | During procedure
  Time from procedure start (insertion of the colonoscope) until colon inspection during a typical withdrawal from cecum to rectosigmoid including any time needed for interventional procedures (biopsies, resection).
Endoscope withdrawal time | During procedure
  Time from deepest point of insertion (cecum) needed for complete inspection of the colon, excluding time spent on therapeutic intervention.

OTHER OUTCOMES:
Adverse events (AEs) | During procedure
  Device-, or procedure-related AEs and Serious AEs (SAEs) reported as incidence (%) and frequency (n).
Non-neoplastic resection rate | During procedure
  Number of patients with no histological confirmation of adenoma, advanced adenoma, SSL, large hyperplastic polyp or carcinoma in any excised lesion divided by the number of colonoscopies where at least one polyp was resected

CONTACTS AND LOCATIONS:
Overall Officials: Karolin Boecker, Study Director — Olympus Europa SE & Co. KG
Locations (6):
- ZU Leuven, Leuven, Belgium
- Germany (2):
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Universitätsklinikum Ulm, Ulm
- Spain (2):
  - Fundación Biomédica Galicia Sur, Pontevedra
  - Hospital Universitari I Politécnic La Fe, Valencia
- Linköping Universitetssjukhus, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No